CLINICAL TRIAL: NCT00004171
Title: Autologous Blood Stem Cell Transplantation in Patients With Hodgkin's Disease and Non-Hodgkin's Lymphoma Who Have Had Prior Radiation Therapy
Brief Title: Peripheral Stem Cell Transplantation Following Radiation Therapy in Treating Patients With Hodgkin's Disease or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 87H6T; NU-87H6T; NCI-G99-1638
Record Dates: First submitted 1999-12-10; First posted 2004-03-01 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; childhood immunoblastic large cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Busulfan; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by peripheral stem cell transplantation in treating patients who have Hodgkin's disease or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and response to intensive chemotherapy followed by autologous peripheral blood stem cell transplantation in patients with Hodgkin's disease or non-Hodgkin's lymphoma who have received prior chemotherapy and/or radiotherapy.

OUTLINE: Patients receive oral busulfan every 6 hours on days -9 to -6 and cyclophosphamide IV over 2 hours on days -5 to -2. Autologous peripheral blood stem cells are reinfused on day 0. Patients are followed monthly for 1 year.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Hodgkin's disease OR Histologically proven non-Hodgkin's lymphoma (NHL) Intermediate grade OR Large cell immunoblastic (high grade) Refractory to standard therapy or relapsed following initial complete remission Must have received radiotherapy to the extent that no longer eligible for involved field radiation, cyclophosphamide, or total body irradiation No CNS disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: Physiologic 65 and under Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: No active heart disease No congestive heart failure No myocardial infarction in the last 3 months No significant arrhythmia requiring medication Pulmonary: No significant nonneoplastic pulmonary disease No chronic obstructive pulmonary disease Diffusing capacity at least 50% predicted OR FEV1 and/or FVC at least 75% predicted (unless due to NHL or Hodgkin's disease) Other: HIV negative No clinical evidence of AIDS

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo I. Gordon, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States